CLINICAL TRIAL: NCT05660980
Title: Phase I/II Study of the Safety, Tolerability, Acceptability, and Pharmacokinetics of Oral and Long-Acting Injectable Cabotegravir and Rilpivirine in Virologically Suppressed Children Living With HIV-1, Two to Less Than 12 Years of Age
Brief Title: Study of Oral and Long-Acting Injectable Cabotegravir and Rilpivirine in Virologically Suppressed Children Living With HIV-1, Two to Less Than 12 Years of Age
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMPAACT 2036; DAIDS Study ID (Other: 38932)
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Cohort 1 will receive Once daily oral CAB + oral RPV through the Week 4b visit, followed by intramuscular injection doses of CAB LA + RPV LA every four weeks (Q4W dosing regimen) or every eight weeks (Q8W dosing regimen)
  Interventions: Drug: Once daily CAB tablet + RPV tablet; Drug: Long acting CAB injectable + long acting RPV injectable
- Cohort 2A (Experimental): Cohort 2A: Once daily doses of oral CAB + oral RPV through the Week 4b visit, followed by Q4W or Q8W intramuscular injection doses of CAB LA + RPV LA.
  Interventions: Drug: Once daily CAB tablet + RPV tablet; Drug: Long acting CAB injectable + long acting RPV injectable
- Cohort 2B (Experimental): Cohort 2B: Q4W or Q8W intramuscular injection doses of CAB LA + RPV LA.
  Interventions: Drug: Long acting CAB injectable + long acting RPV injectable

INTERVENTIONS:
Drug: Once daily CAB tablet + RPV tablet — Tablet
  Arms: Cohort 1; Cohort 2A
Drug: Long acting CAB injectable + long acting RPV injectable — Injectable
  Arms: Cohort 1; Cohort 2A
Drug: Long acting CAB injectable + long acting RPV injectable — Injectable
  Arms: Cohort 2B

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics (PK), safety, tolerability, and acceptability of a long-acting injectable Cabotegravir and Rilpivirine in Virologically Suppressed Children Living with HIV-1, Two to Less Than 12 Years of Age

DETAILED DESCRIPTION:
This is a Phase I/II, multicenter, open-label, non-comparative study to evaluate the safety, tolerability, acceptability, and PK of oral CAB and oral RPV followed by long-acting injectable CAB (CAB LA) and long-acting injectable RPV (RPV LA) to propose the weight-band dosing in virologically suppressed children living with HIV-1 aged two to less than 12 years. The study will also assess the long-acting injectable regimen with and without an oral lead-in period in the same study population.

Following completion of the study, if it is not possible for participants to access injections of CAB LA and RPV LA from non-study sources all participants may enter a Study Safety Extension (SSE) period. During the SSE period ongoing safety information to monitor for toxicities will be collected.

ELIGIBILITY:
Inclusion Criteria, Step 1: Entry for Cohort 1, Cohort 2a, and Cohort 2b

* Parent or legal guardian is willing and able to provide written permission for child's study participation and, when applicable per institutional review board/ethics committee (IRB/EC) policies and procedures, child is willing and able to provide written assent for study participation.

Note: All sites must follow all applicable IRB/EC policies and procedures; for US sites, this includes single IRB (sIRB) policies and procedures.

* Age two years old to less than 12 years old at entry
* Body weight ≥10 kgs and <40 kgs at entry
* At entry, willing and able to comply with the study visit schedule and other study requirements, as determined by the site investigator or designee.
* Confirmed HIV-1-infection based on documented testing of two samples collected from two separate blood collection tubes per Sample #1 and Sample #2 requirements. Test results may be obtained from medical records or from testing performed during the study screening period
* Has been on a stable unchanged ART regimen consisting of two or more drugs from two or more antiretroviral drug classes for at least six consecutive months (defined as 180 consecutive days) prior to entry.
* Has no prior history of switching ART regimens for reasons related to treatment failure based on parent/guardian report and/or available medical records.

Note: Participants undergoing dose modifications for growth or who have switched to a new formulation due to toxicity, tolerability, or changes in national treatment guidelines are considered eligible per this inclusion criterion. Treatment failure should be defined by local guidelines.

* From a specimen collected less than six months (defined as within 179 days) prior to entry, has at least one of the following documented plasma HIV-1 RNA results:

  * <50 copies/mL, or
  * less than the lower limit of detection of the assay
* From a specimen collected in the 6-18 months (defined as 180 to 545 days) prior to entry, has at least one of the following documented plasma HIV-1 RNA results:

  * <50 copies/mL, or
  * less than the lower limit of detection of the assay
* At screening, a documented plasma HIV-1 RNA <50 copies/mL.

Note: HIV-1 RNA test results at screening cannot be used to satisfy previously listed inclusion criterion. If participant does not have a documented HIV-1 RNA test result at screening that satisfies previously listed criteria, they should be referred for standard of care testing and return at a later date for screening.

* Has normal, Grade 1, or Grade 2 results for all the following laboratory tests at screening (i.e., within 28 days prior to entry) based on grading per the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events:

  * AST (<5.0 x ULN)
  * ALT (<5.0 x ULN)
  * Total bilirubin (<2.6 x ULN)
  * Lipase (<3 x ULN)
  * Estimated glomerular filtration rate (eGFR; ≥60 ml/min/1.73 m2)
  * Platelets (≥50,000 cells/mm3 or ≥50.00 x 109 cells/L)
  * Hemoglobin (≥8.5 g/dL or ≥5.25 mmol/L)
  * Neutrophils (≥600 cells/mm3)

Note: Laboratory tests may be repeated during the study screening period (i.e., within 28 days prior to entry), with the latest result used for eligibility determination. ALT and total bilirubin should also be assessed

* Has no evidence of chronic hepatitis B infection based on hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), and hepatitis B surface antibody (HBsAb) testing at screening; any of the following three combinations of test results are acceptable for inclusion:

  * HBsAg negative, HBcAb negative, HBsAb negative
  * HBsAg negative, HBcAb negative, HBsAb positive
  * HBsAg negative, HBcAb positive, HBsAb positive
* At screening, has a mean QTc interval (based upon a triplicate reading) less than or equal to 450 msec based on an electrocardiogram (ECG) automated machine readout or calculated using the Fridericia formula.
* For female participants of childbearing potential, not pregnant based upon negative blood or urine pregnancy test at entry. Childbearing potential is defined as nine years of age or older and:

  * Having reached menarche or
  * Engaging in sexual activity (self-reported) that could lead to pregnancy
* For female participants of childbearing potential who are engaging in sexual activity (self-reported) that could lead to pregnancy, at entry, currently using at least one allowable highly effective method of contraception and agrees to use at least one allowable highly effective method of contraception throughout study participation and for at least 30 days after last oral product use and 48 weeks after last injectable study product use.

Highly effective methods of contraception include:

* Surgical sterilization (i.e., hysterectomy, bilateral oophorectomy, tubal ligation, or salpingectomy)
* Contraceptive intrauterine device or intrauterine system
* Subdermal contraceptive implant
* Progestogen injections
* Combined estrogen and progestogen oral contraceptive pills
* Percutaneous contraceptive patch
* Contraceptive vaginal ring

Inclusion Criteria, Step 2: Continuation for Cohort 1 and Cohort 2a to injection phase

All participants enrolled in Cohort 1 or Cohort 2a will be assessed for eligibility to progress from the oral lead-in phase (Step 1) to the injection phase (Step 2), primarily based on the safety assessments from the Step 1 Week 4a study visit. Clinical assessments conducted prior to administering the first injection at the Week 4b visit will also be used to confirm eligibility to receive the injectable study product.

All of the following criteria must be met in order for a participant enrolled in Cohort 1 or Cohort 2a to be included in Step 2

* Currently enrolled as a participant in Step 1.
* Has normal, Grade 1, or Grade 2 results from all of the following laboratory test results based upon specimens collected at the Week 4a study visit or from confirmatory repeat testing of Week 4a study visit laboratory tests:

  * AST (<5.0 x ULN)
  * ALT (<5.0 x ULN)
  * Lipase (< 3 x ULN)
  * Estimated glomerular filtration rate (eGFR; ≥60 ml/min/1.73 m2))
  * Platelets (≥50,000 cells/mm3 or ≥50.00 x 109 cells/L)
  * Hemoglobin (≥8.5 g/dL or ≥5.25 mmol/L)
  * CK (<10 x ULN)

Note: For a Grade 2 ALT test result from this visit, refer to protocol for required participant management.

* For female participants of childbearing potential not pregnant based upon negative blood or urine pregnancy test at the Week 4b study visit.
* Assessed by the IoR or designee as sufficiently adherent to study products in Step 1 to permit an adequate evaluation of safety and tolerability as part of the oral lead in phase prior to entry into the injection phase.

Inclusion Criteria for Parents/Caregivers

Parents/caregivers of participants will be considered for enrollment to complete quantitative behavioral surveys and/or qualitative in-depth interviews (IDIs), as indicated in the SoE. One parent/caregiver per participant should be enrolled to complete all behavioral assessments, including the IDI, when applicable. Informed consent for parent/caregiver enrollment should be obtained at the entry visit, after the child participant's eligibility has been confirmed, and may be completed at a later date, if necessary. However, parent/caregiver consent must occur prior to any study assessments being conducted. The enrolled caregiver may be the different than the parent or legal guardian who provided written permission for the child to participate. If, at any point the enrolled parent/caregiver for a given participant withdraws from the study or is unable to complete remaining study assessments for any reason, they may be replaced.

Caregivers must meet the following criteria to be eligible to enroll in IMPAACT 2036:

* 18 years of age or older
* Able and willing to provide written informed consent consistent with site IRB/EC policies and procedures
* Caregiver, defined as a biological parent, legal guardian, or other person who provides significant emotional, psychological, and/or physical care to a child enrolled in IMPAACT 2036, based on self-report

Exclusion Criteria, Step 1: Entry for Cohort 1, Cohort 2a, and Cohort 2b

Potential participants must be excluded from the study if any of the conditions specified below are identified during the screening period (i.e., within 28 days prior to study entry). The screening period begins when parental permission and informed assent (if applicable) are obtained and ends immediately prior to enrollment. For criteria involving a potential participant's medical history, it is expected that each exclusionary condition will be assessed at screening and subsequently reviewed and confirmed on the day of study entry, prior to enrollment. In these criteria, "at entry" is used to refer to the day of enrollment in the study

* Within 6 months prior to entry, any HIV-1 RNA value >400 copies/mL OR two consecutive "viral blips," defined as an HIV-1 RNA value ≥50 copies/mL but ≤400 copies/mL.
* As determined by the IoR or designee, and based on available medical records, known or suspected resistance to NNRTIs.

Note: Prior receipt of NNRTIs for prophylaxis or treatment is not exclusionary

* As determined by the IoR or designee, and based on available medical records, known or suspected resistance to INSTIs.
* Ongoing congestive heart failure, symptomatic arrhythmia, or any current clinically significant cardiac disease, as determined by the IoR or designee, and based on available medical records.
* Has any of the following, as determined by the IoR or designee based on participant/parent/guardian report and available medical records:

  * Current hepatitis C infection
  * Current clinically significant hepatic disease
  * Current or anticipated need for chronic anti-coagulation
  * History of known or suspected bleeding disorder, including a history of prolonged bleeding
  * History of sensitivity to heparin or heparin-induced thrombocytopenia, as determined by the IoR or designee, based on available medical records
  * Risk factors for Torsade de Pointes (e.g., heart failure, hypokalemia, hypomagnesemia)
  * Known or suspected allergy to study product components.
  * Known phobia to needles
* More than one seizure within one year (defined as within 365 days) prior to entry, or unstable or poorly controlled seizure disorder, as determined by the IoR or designee, and based on available medical records.
* Has the following combination of laboratory test results at screening (i.e., from specimens collected within 28 days prior to entry): ALT greater than or equal to 3 x ULN and total bilirubin greater than or equal to 1.5 x ULN and direct bilirubin greater than 35% of total bilirubin.
* At entry, known active tuberculosis infection, as determined by the IoR or designee based on participant/parent/guardian report and available medical records.
* At entry, any ongoing pancreatitis as determined by the IoR or designee based on participant/parent/guardian report and available medical records.
* At entry, has symptoms suggestive of active coronavirus disease 2019 (COVID-19) or test results or contacts that require quarantine per local clinical practice, public health, and/or infection control guidelines as determined by the IoR or designee based on participant/parent/guardian report and available medical records.

Note: Potential participants with symptoms suggestive of active COVID-19, test results, and/or contacts that require quarantine may resume screening (or be re-screened) after symptoms have resolved and applicable quarantine requirements have been completed.

* Receipt of any prohibited medication within 7 days prior to entry, with the exception of antiviral agents that are part of the participant's ART regimen, as determined by the site investigator based on participant/parent/guardian report and available medical records

Note: Medications and vaccines approved for emergency use (e.g., COVID vaccines) that do not appear in the IMPAACT 2036 Prohibited and Precautionary Medications listing are not exclusionary may be administered as per standard of care.

* Any past or current exposure to CAB LA or RPV LA
* At entry, based on physical examination, has a current inflammatory skin condition that compromises the safety of intramuscular injections, as determined by the IoR or designee.
* At entry, based on physical examination, has a dermatological condition overlying the buttock or upper thigh region, which, in the IoR or designee's opinion, may interfere with the interpretation of injection site reactions.
* Enrolled in another clinical trial of an investigational agent, device, or vaccine.
* Has any documented or suspected clinically significant medical or psychiatric condition or any other condition or social circumstance that, in the opinion of the site investigator, would make participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Exclusion Criteria, Step 2: Continuation for Cohort 1 and Cohort 2a to injection phase

Participants in Cohort 1 or Cohort 2a who meet any of the following criteria will be excluded from Step 2:

* Has permanently discontinued oral study product.
* Occurrence of any grade 3 or higher adverse event assessed as related to study product during Step 1.
* Any other condition or social circumstance situation that, in the opinion of the IoR or designee, would make continued study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Exclusion Criteria for Parents/Caregivers

* Any condition or social circumstance situation that, in the opinion of the IoR or designee, would make study participation unsafe for the caregiver or the child study participant, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2027-07-27 (Estimated)

PRIMARY OUTCOMES:
AUC (Cohort 1, tablets) | At week 2
  Area under the curve from start of dose to 8 hours post dose
CL/F (Cohort 1, tablets) | At week 2
  apparent clearance from start of dose to 8 hours post dose
Cmax (Cohort 1, tablets) | At week 2
  Peak concentration from start of dose to 8 hours post dose
Tmax (Cohort 1, tablets) | At week 2
  Time of maximal concentration from start of dose to 8 hours post dose
Pre-dose concentrations (C0) (Cohort 1, tablets) | At week 2
Week 5 concentrations (C5WK) (Cohort 1, injections) | Through week5
Week 12 concentrations (C12WK) (Cohort 1, injections) | Through week 12
Trough concentrations (Ct) prior to IM doses through Week 24 (Cohort 1, injections) | Through week 24
Accumulation Ratio at week 24 and week 8 (Cohort 1, injections) | At week 8 and 24
Proportion of children who experience a drug related safety event during the CAB + RPV oral lead-in period (Cohort 1) | Through week 4a
Proportion of children who experience a grade 3 of higher adverse event during the CAB + RPV oral lead-in period (Cohort 1) | Through week 4a
Proportion of children who experience an SAE during the CAB + RPV oral lead-in period (Cohort 1) | Through week 4a
Proportion of children who experience premature permanent discontinuation study treatment due to an adverse event during the CAB + RPV oral lead-in period (Cohort 1) | Through week 4a
Proportion of children who experience a drug-related safety failure event during the 24 weeks of CAB + RPV (oral and injectable) (Cohort 1) | Week 4b through week 28
Proportion of children who experience a grade 3 or higher adverse event during the 24 weeks of CAB + RPV (oral and injectable) (Cohort 1) | Week 4b through week 28
Proportion of children who experience an SAE during the 24 weeks of CAB + RPV (oral and injectable) (Cohort 1) | Week 4b through week 28
Proportion of children who experience premature permanent discontinuation study treatment due to an adverse event during the 24 weeks of CAB + RPV (oral and injectable) (Cohort 1) | Week 4b through week 28

SECONDARY OUTCOMES:
Accumulation ratios Wk 24:Wk 8 and Wk 48: Wk 8 (Cohort 2a), Wk 20:Wk4 and Wk 44: Wk 4 (Cohort 2b | At week 8, 48 and 72
Ct prior to IM doses through Week. 24 and Week. 48 (Cohort 2a) | At Week. 24 and Week. 48
Ct prior to IM doses through Wk. 20 and Wk. 44 (Cohort 2b) | At week 20 and 44
Proportion of children who experience a drug-related safety failure event through Weeks 48 and 72 of CAB + RPV (oral and injectable) (Cohort 1) | Through week 48 and 72
Proportion of children who experience a grade 3 or higher adverse event through Weeks 48 and 72 of CAB + RPV (oral and injectable) (Cohort 1) | Through week 48 and 72
Proportion of children who experience an SAE through Weeks 48 and 72 of CAB + RPV (oral and injectable) (Cohort 1) | Through week 48 and 72
Proportion of children who experience premature permanent discontinuation study treatment due to an adverse event through Weeks 48 and 72 of CAB + RPV (oral and injectable) (Cohort 1) | Through week 48 and 72
Proportion of children who have HIV-1 RNA <50 and ≥50, copies/ml at Weeks 24, 48, and 72 using the FDA Snapshot algorithm (Cohort 1) | At weeks 24, 48 and 72
Proportion of children who have HIV-1 RNA <200 and ≥200 copies/ml at Weeks 24, 48, and 72 using the FDA Snapshot algorithm (Cohort 1) | At weeks 24, 48 and 72
Proportion of children with confirmed virologic failure at Weeks 24, 48 and 72 while on CAB + RPV (Cohort 1) | At weeks 24, 48 and 72
Child and/or parent/caregiver responses to questionnaires about CAB or RPV side effects, pain associated with injections, and injection site reactions at Weeks 24, 48, and 72 (Cohort 1) | At Weeks 24, 48, and 72
Child and/or parent/caregiver reported attitudes about CAB or RPV, including willingness to use at Weeks 24, 48, and 72 (Cohort 1) | At weeks 24, 48 and 72
Proportion of participants who had genotypic and phenotypic resistance to CAB or RPV among children who experience virologic failure while on CAB + RPV (Cohort 1) | Through week 72
Median for CD4 count and percentage at Weeks 24, 48 and 72 (Cohort 1) | At weeks 24, 48 and 72
Median change from baseline CD4 count and percentage at Weeks 24, 48 and 72 (Cohort 1) | At weeks 24, 48 and 72
Child and/or parent/caregiver response to questionnaires (Cohort 2) | at week 44 and 48
  about CAB or RPV side effects, pain associated with injections and injection site reactions for children who are on 48 weeks of CAB+RPV(oral and injectable) OR 44 weeks of CAB LA+RPV LA (injectable)
Child and/or parent/caregiver reported attitudes about CAB (Cohort 2) or RPV, including willingness to use for children who are on 48 weeks of CAB + RPV (oral and injectable) OR 44 weeks of CAB LA + RPV LA (injectable) | At week 44 and 48
Proportion of children who experience a drug-related safety failure event during the 48 weeks of CAB + RPV (oral and injectable) OR the 44 weeks of CAB LA + RPV LA (injectable) (Cohort 2) | At week 44 and 48
Proportion of children who experience a grade 3 or higher adverse event during the 48 weeks of CAB + RPV (oral and injectable) OR the 44 weeks of CAB LA + RPV LA (injectable) (Cohort 2) | At week 44 and 48
Proportion of children who experience an SAE during the 48 weeks of CAB + RPV (oral and injectable) OR the 44 weeks of CAB LA + RPV LA (injectable) (Cohort 2) | At week 44 and 48
Proportion of children who experience premature permanent discontinuation study treatment due to an adverse event during the 48 weeks of CAB + RPV (oral and injectable) OR the 44 weeks of CAB LA + RPV (Cohort 2) LA (injectable) | At week 44 and 48
Proportion of children who have HIV-1 RNA <50 and ≥50, copies/ml using the FDA Snapshot algorithm for children who are on 48 weeks of CAB + RPV (oral and injectable) OR 44 weeks of CAB LA + RPV LA (injectable) (Cohort 2) | At week 44 and 48
Proportion of children who have HIV-1 RNA <200 and ≥200 copies/ml using the FDA Snapshot algorithm for children who are on 48 weeks of CAB + RPV (oral and injectable) OR 44 weeks of CAB LA + RPV LA (injectable) (Cohort 2) | At week 44 and 48
Proportion of children with confirmed virologic failure while on treatment for children who are on 48 weeks of CAB + RPV (oral and injectable) OR 44 weeks of CAB LA + RPV LA (injectable) (Cohort 2) | At week 44 and 48
Median and Interquartile Range for CD4 count and percentage for children who are on 48 weeks of CAB + RPV (oral and injectable) OR 44 weeks of CAB LA + RPV LA (injectable) (Cohort 2) | At week 44 and 48
Median and Interquartile Range change from baseline CD4 count and percentage for children who are on 48 weeks of CAB + RPV (oral and injectable) OR 44 weeks of CAB LA + RPV LA (injectable) (Cohort 2) | At week 44 and 48
Proportion of participants who had genotypic and phenotypic resistance to CAB and RPV among children who experience virologic failure while on 48 weeks of CAB + RPV (oral and injectable) OR while on 44 weeks of CAB LA + RPV LA (injectable) (Cohort 2) | At week 44 and 48
LA dosing: Ct prior to IM doses at Wk. 48 and Wk. 72 and accumulation ratios (Wk. 48:Wk. 8 and Wk. 72:Wk. 8) (Cohort 1) | At week 8 and 48

OTHER OUTCOMES:
CAB and RPV concentrations 8 to 48 weeks following final IM dose | At week 8 and 48
Proportion of children who experience a drug-related safety failure event through 48 weeks following permanent discontinuation of CAB LA + RPV LA | Through week 48
Proportion of children who experience a grade 3 or higher adverse event through 48 weeks following permanent discontinuation of CAB LA + RPV LA | Through week 48
Proportion of children who experience an SAE through 48 weeks following permanent discontinuation of CAB LA + RPV LA | Through week 48
PO dosing: Wk. 2 AUC, CL/F, Cmax, Tmax, and pre-dose concentrations (C0) by administration mode | At week 2

CONTACTS AND LOCATIONS:
Locations (12):
- United States (2):
  - Site 5030, Emory University School of Medicine NICHD CRS, Atlanta, Georgia
  - Site 6501, St. Jude Children's Research Hospital CRS, Memphis, Tennessee
- Botswana (2):
  - Site 12701, Gaborone CRS, Gaborone
  - Site 12702, Molepolole CRS, Gaborone
- Brazil (2):
  - Site 5073, SOM Federal University Minas Gerais Brazil NICHD CRS, Belo Horizonte
  - CRS 5071, Instituto de Puericultura e Pediatria Martagao Gesteira Clinical Research Site, Rio de Janeiro
- South Africa (3):
  - Site 30300 Umlazi CRS Site, Umlazi, KwaZulu-Natal
  - Site 8051, Wits RHI Shandukani Research Centre CRS, Johannesburg
  - CRS 8052, Soweto IMPAACT, Johannesburg
- Thailand (3):
  - Siriraj Hospital, Mahidol University NICHD CRS (Site #5115), Bangkok, Bangkoknoi
  - CRS 31784, Chiang Mai University HIV Treatment CRS, Chiang Mai
  - Site 5116, PHPT-Chiangrai Prachanukroh Hospital NICHD CRS, Chiang Rai

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: With whom?
  * Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses?
  * To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available?
  * Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https:// www.impaactnetwork.org/ resources/study-proposals.htm. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.